CLINICAL TRIAL: NCT02533609
Title: Elimination of Antibiotics During Citrate-anticoagulated Continuous-veno-venous-haemodialysis
Acronym: DIADSORBMAB
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Principal Investigator, Klinik für Anästhesiologie, Prof. Dr. D. Kindgen-Milles, Heinrich-Heine University, Duesseldorf
Other Study IDs: 2015-02-ENDVERSION
Record Dates: First submitted 2015-08-20; First posted 2015-08-27 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Acute Kidney Injury; Bacterial Infection
MeSH Terms: conditions — Acute Kidney Injury; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Piperacillin/Tazobactam: Patients undergoing continuous veno-venous renal replacement therapy and treated with this antibiotics
- Imipenem/Cilastatin: Patients undergoing continuous veno-venous renal replacement therapy and treated with this antibiotics

SUMMARY:
Acute kidney injury (AKI) requiring renal replacement therapy is common in critically ill patients. The major causes of AKI are severe sepsis and septic shock requiring effective antibiotic treatment. Patients with sepsis on ICUs usually are haemodynamically instable so that renal replacement therapy is applied using continuous techniques. In recent years, the efficacy of renal replacement therapies has improved, namely by using regional citrate anticoagulation which improves filter lifetime and filter patency. At present, the extent of removal of antibiotic drugs using citrate-anticoagulated CVVHD in critically ill patients has not been investigated thoroughly. Thus, the investigators want to investigate

1. whether and to what extent antibiotic drugs (piperacillin/tazobactam and imipenem/cilastatin) are removed during citrate-anticoagulated CVVHD per se
2. whether filter patency during citrate-anticoagulated CVVD remains stable during a treatment period of 72 h

ELIGIBILITY:
Inclusion Criteria:

* Intensive care patients with acute kidney injury requiring continous renal replacement therapy with citrate-anticoagulation
* Age > 18 y

Exclusion Criteria:

* < 18 y
* Pregnancy
* Contraindications against citrate-anticoagulation or continous renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients with acute kidney injury requiring continous renal replacement therapy with citrate-anticoagulation
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Removal of antibiotic drugs during day 1 - 2 - 3 of citrate anticoagulated CVVHD (mg/d) | up to three days
  Total hemofilter clearance (ml/min) of imipenem/cilastatin and piperacillin/tazobactam on each treatment day during an 8-hour dosing interval using blood sided clearance
  - Total amount of antibiotic drug which is eliminated via the filter during 24 h using filter clearance and delivered dialysis dose during 24 h
Filter patency during day 1 - 2 - 3 of citrate anticoagulated CVVHD | up to three days
  Filter patency is calculated as a function of the sieving coefficient for small solutes (i.e. creatinine and the respective antibiotic drugs) over the first 72 h, Sieving coefficient is without dimension

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Kindgen-Milles, Prof., Study Director — Department of Anesthesiology
Locations (1):
- Prof. Kindgen-Milles, Düsseldorf, Germany